CLINICAL TRIAL: NCT02563730
Title: Open Label Trial of Utility of Cryobiopsy in the Multidisciplinary Diagnosis of Idiopathic Interstitial Lung Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Boeckeler, Michael, MD, University Hospital Tuebingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CRYO-VATS
Record Dates: First submitted 2015-05-02; First posted 2015-09-30 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Interstitial Lung Disease
Keywords: Cryobiopsy; lung biopsy; interstitial lung disease
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lung biopsy (Experimental): assess the additional diagnostic value of cryobiopsy in patients with suspected Idiopathic Interstitial Pneumonia (IIP). Cryoprobe vs VATS
  Interventions: Procedure: Lung biopsy

INTERVENTIONS:
Procedure: Lung biopsy — transbronchial lung biopsy. First kryobiopsy, second open biopsy

SUMMARY:
A multicenter, multinational, prospective study to clarify, whether the addition of cryobiopsy can avoid surgical lung biopsy in a clinically relevant proportion of patients with suspected Idiopathic Interstitial Pneumonia

ELIGIBILITY:
Inclusion Criteria:

* IIP suspected on clinical and radiologic grounds

Exclusion Criteria:

* Age >80y and <18y
* FVC< 55%, DCO<35%
* Platelet count <100000/µl
* acetylsalicylic acid, clopidogrel or equivalent during the last 5 days
* INR > l,3,
* elevated PTT (> 40 s)
* documented pulmonary hypertension PAPS >50mmHg
* HR-CT highly suspicious for sarcoidosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of conclusive diagnosis after bronchoscopy with transbronchial cryobiopsy | two weeks

SECONDARY OUTCOMES:
numer of bleeding events | 1 day
Rate of pneumothoraxes | 1 day
numer of exacerbations after biopsy | 6 weeks
Contribution of BAL and cryobiopsy to diagnosis | 2 weeks
Size of specimen | 2 weeks
Quality of specimen | 2 weeks
Distribution of histological changes in the specimen | 2 weeks
Influence of the size of the cryoprobe in the primary endpoint | 2 weeks
Comparative group (out of trial) - who are referred for VATS directly ['positive control group'] | 6 weeks
Rate of exacerbations after cryobiopsy and after surgical biopsy | 6 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- Germany (3):
  - Ruhrlandklinik, Essen
  - Thoraxklinik, Heidelberg
  - University Hospital Tuebingen, Tübingen
- Ospedale G.B. Morgagni, Forlì, Italy
- Respiratory Department Hospital of Santa Creu i Sant Pau, Barcelona, Spain
- Royal Brompton Hospital, London, United Kingdom